CLINICAL TRIAL: NCT02470689
Title: Diacerin for the Treatment of Epidermolysis Bullosa Simplex
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Head of Division of Research and Development, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TASMC-15-SE-135-14-CTIL
Record Dates: First submitted 2015-05-27; First posted 2015-06-12 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-05

CONDITIONS: Epidermolysis Bullosa Simplex
MeSH Terms: conditions — Epidermolysis Bullosa Simplex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diacerin cream 1% (Active Comparator)
  Interventions: Drug: Diacerin cream
- ultraphil cream (Placebo Comparator)
  Interventions: Drug: Diacerin cream

INTERVENTIONS:
Drug: Diacerin cream — Diacerin tablet solubule in ultraphil cream

SUMMARY:
Epidermolysis bullosa simplex type Dowling-Meara (EBS-DM) is one of the most severe subtypes of EBS. Blisters and erosions of the skin and mucous membranes upon minor trauma are the consequence of dominantly inherited mutations in either the keratin 5 (K5) or keratin 14 (K14) gene, which encode proteins constituting the intermediate filament (IF) network in basal keratinocytes . Autosomal dominant mutations lead to a conformational change and an increased self-aggregation of the protein. Upon stress, aggregates present in the periphery of the cytoplasm, subsequently leading to the disintegration and collapse of the IF network. Clinically, patients suffer from blistering of the skin and mucous membranes upon minor trauma, resulting in an impaired life quality due to pain and pruritus . In vitro studies on Dowling-Meara keratinocytes revealed a significant upregulation of the pro-inflammatory cytokine interleukin-1beta (IL-1ß). Apart from paracrine effects of IL-1ß upon wounding (e.g. attraction of lymphocytes, activation of dermal fibroblasts), IL-1ß also activates keratinocytes via the cjun N-terminal kinase (JNK) stress pathway. The activation of this pathway leads to the activation of a number of transcription factors and the enhanced transcription of a number of genes, like matrix metalloproteinases, kallikreins, but also IL-1ß itself and K14 . Interestingly, this state of activation is constitutive and was also found in keratinocytes from non-lesional sites. It seems that the upregulation of IL-1ß and K14 in the presence of dominant Dowling-Meara mutations, results in a positive feedback loop, potentially aggravating the EBS-DM phenotype. This was strongly corroborated by the fact that when impairing IL1ß signaling, using IL-1ß neutralizing antibody (IL-1Ab) or the small molecule diacerein, expression levels of IL-1ß and K14 decreased and keratinocytes were much less susceptible to heat shock in vitro . Furthermore, activation levels of JNK widely correlated with expression levels of K14 and IL-1ß. (Wally V et al, 2013). These findings led to the hypothesis that blocking IL-1ß will also lead to an amelioration of the EBSDM phenotype in effected patients. Based on previous in vitro findings diacerein was chosen to be topically applied in a pilot study with five patients suffering from EBS-DM. In that study , each participant received 1% diacerein-cream for one armpit, and placebo for the other (randomized withdrawal). The number of blisters was reduced significantly (left: -78%; right: -66% of baseline) within two weeks and remained significantly below the initial level even during withdrawal in four patients. These findings pointed to a relevant effect of diacerein and provide important information for our confirmative study.

Diacerein is a component of the rhubarb root, which is reported to block the release of active IL-1b by inhibiting plasma membrane-bound IL-1 converting enzyme . Diacerien is already approved for systemic application in osteoarthritis . In general, small molecules (SM) are low molecular weight compounds with biological functions that can influence molecular processes. They allow a symptomatic treatment, offering a short-term benefit for patients in terms of an amelioration of the phenotype. Although this kind of treatment does not correct genetic alterations, it can still be highly beneficial by damping down disease symptoms, thereby increasing life quality and minimizing secondary manifestations.

It is important to emphasize that besides dressings, there are currently no other treatments, therefore, investigators do not prevent an accepted treatment for the patient and there is no risk for the participant. The treatment will be given only to the armpits although the disease can involve other areas, so stopping dressings in the armpits during the study does not risk the patient. Should there be any deterioration of the patient, whether it is related to the treatment with diacerein or not, investigators will stop the use of diacerein.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of EBS-DM
2. An age between 6 - 19

Exclusion Criteria:

1. Lack of mutation analysis
2. Intolerance to a component of the cream
3. Pregnancy or Lactation
4. Contemporaneous participation in another clinical trial

Ages: 6 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of blisters | 4 weeks

SECONDARY OUTCOMES:
Number of blisters | 3 months period

CONTACTS AND LOCATIONS:
Overall Officials: Eli Sprecher, Prof., Principal Investigator — Head of Dermatology Department, Ichilov medical center